CLINICAL TRIAL: NCT01500265
Title: Assessment and Monitoring of Renal Proximal Tubular Tolerance of Nucleoside and Nucleotide Analogues Using Early Screening Tools in Patients Chronically Mono-infected With Hepatitis B Virus.
Acronym: HBVSECURE
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I10006 HBVSECURE
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Hepatitis B; Renal Failure With Tubular Necrosis
Keywords: hepatitis B virus; early screening tools; renal proximal tubular tolerance
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and urine samples for determination of TMPi / GFR and FEUA A sample of genomic DNA will be collected after informed consent of the patient from a saliva sample (Saliva autocollection kits) in order to investigate genetic polymorphism in transporters responsible for the renal elimination of TDF and ETV.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patient naive: Patient with hepatitis B virus naive untreated
  Interventions: Biological: plasma and urine samples, sample with ADN
- Patient with TDF: Patient with hepatits B treated with Tenofovir
  Interventions: Biological: plasma and urine samples, sample with ADN
- Patient with ETV: Patient with hepatitis B virus treated with Entecavir
  Interventions: Biological: plasma and urine samples, sample with ADN

INTERVENTIONS:
Biological: plasma and urine samples, sample with ADN — plasma and urine samples every three months Sample with ADN at baseline

SUMMARY:
Nucleotide analogues are associated in the long term with a risk of proximal tubular nephropathy (PT) with loss of phosphate, and, when compensatory mechanisms are overwhelmed, with osteopenia or osteoporosis. This toxicity has been particularly documented for tenofovir (TDF) in HIV disease, but its prevalence varies widely in the literature and is mainly associated with comorbidities: on average this prevalence is 0.39% after 48 weeks with exceptional cases of Fanconi syndrome described. In HBV monoinfection after 60 months of treatment with TDF, an 11% decrease of creatinine clearance (CreatCl) is observed. A single study showed a significant increase in creatinine level with entecavir (ETV) therapy, a second-generation nucleoside, hitherto not described as nephrotoxic. Furthermore, if the direct renal toxic effect characteristic of HIV in the kidney is well known, the role of HBV is less clear. Thus, HBV treatment appears to have a renal protective effect. The monitoring tools recommended by the SPC, CreatCl and plasma phosphorus level are late markers of tubular damage. The threshold of phosphate tubular reabsorption (TmPi/GFR) and the fractional excretion of uric acid (FEUA) are unexpensive early screening tools. However, the long-term evolution of this subclinical tubular involvement in HBV monoinfection is not known.

DETAILED DESCRIPTION:
260 naive untreated patients, 220 patients treated with TDF and 220 patients treated with ETV and consecutively recruited in this interventional study, will have at baseline and every three months, a determination of phosphorus, creatinine, uric acid in plasma and urine samples for determination of TMPi / GFR and FEUA, and an evaluation of urinary calcium level. Depending on local opportunities, every six months, a urine sample will be stored in a declared biological collection to perform β2-microglobuline and cystatin dosage. A 25-OHD3 and PTH dosage will be conducted annually. A sample of genomic DNA will be collected after informed consent of the patient from a saliva sample (Saliva autocollection kits) in order to investigate genetic polymorphism in transporters responsible for the renal elimination of TDF and ETV. A serum sample will be stored at baseline, at one year and at endpoint for the retrospective dosage of bone markers (bone PAlk, PINP and CTX).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with chronic HBV virus monoinfected
* For groups of patients treated: Patients with an indication of ETV or TDF
* For the group of naive patients: treatment-naive patients who have no indication of treatment (or do not want) for the duration of the study
* globular filtration rate (GFR) ≥ 50 ml / min / 1.73 m2 with no known cause of renal disease
* Patients who have given their informed and written informed consent
* Women of childbearing potential with an effective method of contraception without interruption for the duration of the research and during the 4 months after stopping treatment

Exclusion Criteria:

* Patients co-infected with HIV, hepatitis C or hepatitis Delta
* Patients who have already received the TDF in the group to receive the TDF and having already received ETV in the group to receive ETV
* Patient with a GFR <50 ml / min / 1.73 m2 or with known causes of renal disease
* Patient with hypophosphatemia <0.48 mmol / l
* Patients with hepatocellular carcinoma (diagnosed or suspected)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with hepatitis B virus
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
the prevalence of "subclinical" proximal tubular abnormalities | 2 years
  to compare at 2 years the prevalence of "subclinical" proximal tubular abnormalities (TmPi/GFR and FEUA) in 3 groups of HBV monoinfected patients treated with TDF, ETV or untreated.

SECONDARY OUTCOMES:
the prevalence at baseline of "subclinical" proximal tubular abnormalities | 1 day
  to describe the prevalence at baseline, and the cumulative incidence of these abnormalities during the follow-up and determine the proportion of patients who present at 2 years an impaired CreatCl, an hypophosphatemia and an hypercalciuria (suggesting a bone impact), according to the presence or absence of "subclinical" proximal tubular abnormalities.

CONTACTS AND LOCATIONS:
Locations (25):
- France (25):
  - CHU d'Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Besancon, Besançon
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux
  - CHU de Brest, Brest
  - CHU de CAEN, Caen
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - AP-HP - Hôpital Beaujon, Clichy
  - Centre Hospitalier Laennec de Creil, Creil
  - Centre Hospitalier d'Hyères, Hyères
  - Centre Hospitalier de La Roche sur Yon, La Roche-sur-Yon
  - AP-HP - Hôpital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lille - Hôpital Huriet, Lille
  - CHU de Limoges - Fédération Hépatologie, Limoges
  - Hospices Civils de Lyon - Hôpital Croix Rousse, Lyon
  - CHU de Montpellier - Hôpital Saint Eloi, Montpellier
  - CHU de Nice, Nice
  - AP-HP - Hôpital La Pitié Salpétrière, Paris
  - AP-HP - Hôpital Bichat, Paris
  - CHU de Bordeaux - Hôpital Haut Levêque, Pessac
  - CHU de Point à Pitre, Point À Pitre
  - CHU de Poitiers, Poitiers
  - CHU de Strasbourg - Hôpital Civil, Strasbourg
  - CHU de Tours - Hôpital Trousseau, Tours
  - CHU de Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy